CLINICAL TRIAL: NCT02866474
Title: Efficacy of the Implementation of a Food and Nutritional Support Strategy Adapted to Dependent Elderly Subjects: Controlled Trial.
Brief Title: Efficacy of the Implementation of a Food and Nutritional Support Strategy Adapted to Dependent Elderly Subjects
Acronym: RENES+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: VVW ancillaireANR 2013
Record Dates: First submitted 2016-08-10; First posted 2016-08-15 (Estimated); Last update posted 2024-02-12 (Actual); Status verified 2018-06

CONDITIONS: Nutrition; Elderly
MeSH Terms: interventions — Food Services

ARMS (2):
- - Puteaux or Paris for elderly persons (Other)
  Interventions: Dietary Supplement: population living at home with meals on wheels
- -Two EHPAD in Lyon for elderly persons living (Other)
  Interventions: Dietary Supplement: population living in an EHPAD

INTERVENTIONS:
Dietary Supplement: population living at home with meals on wheels
  Arms: - Puteaux or Paris for elderly persons
Dietary Supplement: population living in an EHPAD
  Arms: -Two EHPAD in Lyon for elderly persons living

SUMMARY:
Malnutrition particularly affects people who delegate the preparation of their meals with 46% of persons living at home and using a meals-on-wheels service, or those in old people's homes (Etablissement d'Hebergement pour Personnes Agees Dependantes - EHPAD) at risk of malnutrition, compared with 16% in persons who have help, but not for their meals, and 8% in independent persons (Aupalesens Survey). This proportion, which is particularly high, is essentially due to the absence or insufficient level of individual monitoring of the nutritional status of these "dependent" populations despite the different recommendations. EHPAD (old people's homes) are invited to respect meal rhythms, to adapt the nutritional and gustatory qualities of the food, to propose a pleasant environment (Survey CLCV 2012: data collection in 2012); in parallel, few professionals are really trained in the needs of the elderly. In meals-on-wheels services, apart from the distribution of meals, no nutritional follow-up is proposed (Guide 2012).

Symmetrically, the constant search to control costs in western healthcare systems has led managers to systematically reduce care costs, in particular those that are not directly related to medico-pharmaceutical or care personnel expenditure in the strictest sense. In the collective catering services, there is, for example, a systematic effort to reduce daily "costs/materials", without measuring the global cost related to the efficacy of care.

The present work is part of the RENESSENS project: these studies will be conducted in two elderly populations, one living at home and receiving meals on wheels daily and a regular visit of a dietician, who will propose individual nutritional follow-up and the second living in an old people's home (EHPAD) that will benefit from the improved management of its catering service (good culinary practices, including specific training for personnel and meals adapted to the needs of residents). The principal aim of these two studies will be common and will be to evaluate the efficacy of this specific type of management of meals and nutrition compared with a reference meals-on-wheels service and a reference EHPAD.

ELIGIBILITY:
Inclusion Criteria:

* persons or their persons of trust who have given oral consent
* Age ≥ 65 years
* Persons living at home using a meals on wheels service every day or living in an old people's home (EHPAD)

Exclusion Criteria:

* Persons without national health insurance cover
* Persons requiring enteral or parenteral nutrition
* Persons in an exclusion period for a previous study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2018-03-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the nutritional status via the evolution of the Mini Nutritional Assessment (MNA) score including the evolution of weight | Change with regard to Day 0, at three months , at six months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France